CLINICAL TRIAL: NCT06361615
Title: Effect of a Dual-task Intervention Program on Physical and Cognitive Function in Institutionalized Older Adults: a Randomized Clinical Trial
Brief Title: Effect of a Dual-task Intervention Program on Physical and Cognitive Function
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Americas (Other)
Responsible Party: Principal Investigator, Ignacio Astudillo Ganora, Principal Investigator, University of Americas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEC_FP_2023042
Record Dates: First submitted 2024-04-05; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Functional Movement Disorder; Fragility
Keywords: dual task exercise; institutionalized; physical function
MeSH Terms: conditions — Conversion Disorder

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: Although blinding is not possible for participants in exercise-intervention research, the outcome assessors and data analysts were masked to group assignments. The study was unblinded after the statistical analyses were completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simple-Task (multicomponent physical exercise) (Active Comparator): Single-task (ST) training group developed an exercise program based on Functional Exercise Circuit (FEC) protocol
  Interventions: Other: Single-Task
- Dual-Task training (multicomponent physical exercise + cognitive tasks) (Experimental): Dual-task (DT) training group performed motor (FEC) plus cognitive tasks
  Interventions: Other: Dual-Task

INTERVENTIONS:
Other: Single-Task — Single-task (ST) training group developed an exercise program based on Functional Exercise Circuit (FEC) protocol. This exercise program has been published previously12, which considered 15 different exercises in a functional exercise circuit.
  Arms: Simple-Task (multicomponent physical exercise)
Other: Dual-Task — DT training (multicomponent physical exercise + cognitive tasks)
  Arms: Dual-Task training (multicomponent physical exercise + cognitive tasks)

SUMMARY:
Aim: to compare the effects of single-task (ST) and dual-task (DT) training on physical and cognitive function in institutionalized older adults in 1 month.

Methods: Participants were assigned randomly into two groups, ST (multicomponent physical exercise) and DT training (multicomponent physical exercise + cognitive tasks). Both groups performed the exercise three times per week for 1 month. Short Physical Performance Battery (SPPB), handgrip strength, Barthel Index and Montreal Cognitive Assessment (MoCA) were used to assess physical and cognitive performance, respectively. Variables were measured at the beginning (V1),at the end of the exercise (V2), as well as one month later (V3). Paired Student's t-test and lineal logistic regressions models were used to explore the effect of the exercise interventions.

ELIGIBILITY:
Inclusion Criteria:

* Institutionalized older people between 65 and 75
* mild to moderate cognitive impairment

Exclusion Criteria:

* Acute or chronic pathologies that prevent exercise

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-04-05 (Estimated)

PRIMARY OUTCOMES:
Short Physical Performance Battery (SPPB) | 4 weeks
  The SPPB is a battery of tests that include: the 4-meter walking test (4MWT) performed at usual pace, the 5-times sit-to-stand test (5STS), and Romberg balance test, assessing the ability of standing upright in three progressively standing conditions (feet together, semi-tandem and full-tandem) for a maximum period of ten seconds. SPPB scores range from 0 (inability to complete the test) to 4 (best performance), obtaining a total score ranging from 0 (worst performance) to 12 (best performance)14.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | 4 weeks
  MoCA15 was used to assess cognitive status. This test evaluates older adults' attention, language, calculation, orientation, construction, visual and memory. This test has been validated in Spanish16and has cut-off scores adjusted to the Chilean population17. maximum score is 30 points, where 26 points or more is considered normal
Barthel Index | 4 weeks
  Disability status was assessed by the Barthel Index18. This test measures the individual's independence in Basic Activities of Daily Living (BADLs). Barthel Index classifies individuals in four categories: severe disability (scores from 0 to 60), moderate disability (scores from 65 to 85), mild disability (from 90 to 95) and no disability (scores of 100).
Isometric Handgrip Strength (IHS) | 4 weeks
  IHS in both hands were evaluated by using a hydraulic JAMAR dynamometer (J. A. Preston Corporation, Clifton, NJ, USA) following standard procedures19. The best of two performances with one minute of resting between them was registered.
Immobility Syndrome Scale | 4 weeks
  Staging of dismobility was assessed by the tool proposed by Dinamarca (ETADI) 20. ETADI tries to classify older individuals according to their immobility level: stage 1 corresponds to the level in which the patient can spend most of the day in standing, stage 2, sedentary, and stages 3, 4 and 5 correspond to the substages of bed rest. Sub-stage "A" is related to greater independence and "B" to greater dependence on the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de las Americas, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No